CLINICAL TRIAL: NCT00818519
Title: A Multicenter, Double-blind, Randomized, Placebo Controlled Study to Evaluate the Efficacy and Safety of an Oral Contraceptive Preparation YAZ (Drospirenone 3 mg / Ethinylestradiol 20 µg) for 6 Treatment Cycles in Women With Moderate Acne
Brief Title: GA YAZ ACNE in China Phase III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91772; 311963 (Other: Company internal); 2014-004612-10 (EudraCT Number)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2011-06-09 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Acne Vulgaris
Keywords: Moderate Acne Vulgaris; Oral contraceptive; Female
MeSH Terms: conditions — Acne Vulgaris | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EE20/Drospirenone (YAZ, BAY86-5300) (Experimental): In the active treatment group, participants received 24 consecutive days of active tablets followed by 4 consecutive days of inactive tablets. The active tablet contained 3 mg DRSP (Drospirenone) and 20µg EE (Ethinyl estradiol).
  Interventions: Drug: EE20/Drospirenone (YAZ, BAY86-5300)
- Placebo (Placebo Comparator): The participants of the placebo group received inert but identical-appearing, color-matched tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EE20/Drospirenone (YAZ, BAY86-5300) — 20µg ethinylestradiol, 3mg drospirenone, tablet, orally, opd
  Arms: EE20/Drospirenone (YAZ, BAY86-5300)
Drug: Placebo — Inert tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of YAZ (drospirenone 3 mg / ethinylestradiol 20 µg) in comparison with placebo in female patients with moderate acne vulgaris over 6 treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women of age 14-45 years
* >1 year post-menarche with moderate acne vulgaris who have no known contraindications to combined oral contraceptives
* Otherwise healthy, except for the presence of moderate acne
* Smokers up to a maximum age of 30 (inclusive) at inclusion

Exclusion Criteria:

* Pregnancy, lactation (less than three menstrual cycles since delivery, abortion, or lactation before start of treatment)
* Obesity (Body Mass Index > 30 kg/m2)
* Hypersensitivity to any ingredient of the study drug
* Any disease or condition that may worsen under hormonal treatment

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 179 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- China (6):
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Chengdu, Sichuan
  - Beijing
  - Shanghai

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Analyzed: 179 participants randomized, 173 in the FAS (Full Analysis Set): 87 in YAZ, 86 in placebo groups, 143 in the PPS (Per Protocol Set): 74 in YAZ, 69 in placebo groups
Pre-assignment Details: 193 participants screened, 14 failed screening: withdrawal of consent (7), inclusion/exclusion criteria not met (6), participant lost/no further information available (1). study drug intake was unknown (3) and 3 participants to whom study drug was never administered (withdrawal of consent or lost to follow-up) were excluded from FAS.
Period: Overall Study
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Started | 89 (2 excluded from FAS because study drug intake unknown or never administered) | 90 (4 excluded from FAS because study drug intake unknown or never administered)
Participants Received Treatment | 87 (= Baseline) | 86 (= Baseline)
Completed | 75 | 71
Not Completed | 14 | 19
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 4 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 4 | 9
Not completed — participant recovered completely | 1 | 0
Not completed — participant will leave for long tme | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of participants was derived from birth date entered onto CRF (Case Report Form)
  Years | 24.0 (5.8) | 23.4 (5.4) | 23.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Cycle 6 to Baseline in the Total Lesion Count (Open and Closed Comedones, Papules, Pustules, and Nodules) in the FAS (Full Analysis Set)
Description: Acne lesions were counted by the trained designee over the entire face. All types of lesions were to be identified and separately counted, i.e., non-inflammatory open and closed comedones, and inflammatory papules, pustules, and nodules. The percent change from Cycle 6 to Baseline was calculated as (total lesion count at Baseline - total lesion count at Cycle 6)/(total lesion count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 87 | 86
Percent change | 66.79 (31.45) | 37.71 (118.73)

2. Primary Outcome: Percent Change From Cycle 6 to Baseline in the Total Lesion Count (Open and Closed Comedones, Papules, Pustules, and Nodules) in the PPS (Per Protocol Set)
Description: as for outcome 1
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: PPS
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 74 | 69
Percent change | 72.63 (27.45) | 55.56 (32.50)

3. Secondary Outcome: Percentage of Participants Classified as "0" or "1" on the 6-point ISGA (Investigator Static Global Assessment) Scale at Screening Visit
Description: ISGA scale 0: Normal, clear skin with no evidence of acne vulgaris; 1: Skin is almost clear: few non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving, not pink-red), no nodular lesions; 2: Few inflammatory lesions, little inflammation, some comedones, no nodular lesions; 3: Non-inflammatory lesions predominate, several inflammatory lesions, one small nodular lesion maybe present; 4: Many inflammatory lesions, up to many comedones, up to a few nodular lesions; 5: Numerous highly inflammatory lesions predominate, many papules and pustules or nodular lesions
Time Frame: Screening visit
Population: Full analysis set at screening
Measure: Number; unit: Percentage of participants
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 87 | 86
Percentage of participants | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants Classified as "0" or "1" on the 6-point ISGA (Investigator Static Global Assessment) Scale at Cycle 1
Description: as for outcome 3
Time Frame: Cycle 1 (Day 15±3 days of Treatment Cycle 1)
Population: FAS, all participants with data for Cycle 1
Measure: Number; unit: Percentage of participants
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 84 | 84
Percentage of participants | 1.2 | 0.0

5. Secondary Outcome: Percentage of Participants Classified as "0" or "1" on the 6-point ISGA (Investigator Static Global Assessment) Scale at Cycle 3
Description: as for outcome 3
Time Frame: Cycle 3 (Day 15±3 days of Treatment Cycle 3)
Population: FAS, all participants with data for Cycle 3
Measure: Number; unit: Percentage of participants
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 81 | 81
Percentage of participants | 2.5 | 4.9

6. Secondary Outcome: Percentage of Participants Classified as "0" or "1" on the 6-point ISGA (Investigator Static Global Assessment) Scale at Cycle 6
Description: as for outcome 3
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6)
Population: FAS, all participants with data for Cycle 6
Measure: Number; unit: Percentage of participants
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 73 | 71
Percentage of participants | 49.3 | 18.3

7. Secondary Outcome: Percent Change From Cycle 6 to Baseline in Inflammatory Lesion Count (Papules, Pustules, and Nodules), Non-inflammatory Lesion Count
Description: Acne lesions were counted by the trained designee over the entire face. All types of lesions were to be identified and separately counted, i.e., non-inflammatory open and closed comedones, and inflammatory papules, pustules, and nodules. The percent change from Cycle 6 to Baseline was calculated as (lesion count at Baseline - lesion count at Cycle 6)/(lesion count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 75 | 71
Percent change
  Inflammatory lesion count | 75.49 (28.11) | 60.88 (29.92)
  Non-inflammatory lesion count | 69.27 (33.75) | 50.24 (49.93)

8. Secondary Outcome: Percent Change From Cycle 6 to Baseline in Lesion Count of Papules
Description: Acne lesions were counted by the trained designee over the entire face. All papules were to be identified and separately counted. The percent change from Cycle 6 to Baseline was calculated as (papule count at Baseline - papule count at Cycle 6)/(papule count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 75 | 71
Percent change | 72.36 (31.32) | 55.03 (40.19)

9. Secondary Outcome: Percent Change From Cycle 6 to Baseline in Lesion Count of Pustules
Description: Acne lesions were counted by the trained designee over the entire face. All pustules were to be identified and separately counted. The percent change from Cycle 6 to Baseline was calculated as (pustule count at Baseline - pustule count at Cycle 6)/(pustule count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 64 | 61
Percent change | 79.88 (40.83) | 78.15 (34.37)

10. Secondary Outcome: Percent Change From Cycle 6 to Baseline in Lesion Count of Nodules
Description: Acne lesions were counted by the trained designee over the entire face. All nodules were to be identified and separately counted. The percent change from Cycle 6 to Baseline was calculated as (nodule count at Baseline - nodule count at Cycle 6)/(nodule count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 32 | 30
Percent change | 95.83 (18.45) | 95.00 (20.13)

11. Secondary Outcome: Percent Change From Cycle 6 to Baseline in Lesion Count of Open Comedones
Description: Acne lesions were counted by the trained designee over the entire face. All open comedones were to be identified and separately counted. The percent change from Cycle 6 to Baseline was calculated as (open comedone count at Baseline -open comedone count at Cycle 6)/(open comedone count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 72 | 69
Percent change | 24.03 (289.46) | 38.31 (94.52)

12. Secondary Outcome: Percent Change From Cycle 6 to Baseline in Lesion Count of Closed Comedones
Description: Acne lesions were counted by the trained designee over the entire face. All closed comedones were to be identified and separately counted. The percent change from Cycle 6 to Baseline was calculated as (closed comedone count at Baseline - closed comedone count at Cycle 6)/(closed comedone count at Baseline)*100, so that improvement is indicated by a larger percent change.
Time Frame: Cycle 6 (Day 15±3 days of Treatment Cycle 6) and Baseline
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 75 | 70
Percent change | 69.52 (42.24) | 48.73 (61.16)

13. Secondary Outcome: Percentage of Participants Classified as "Improved" According to the Investigator's Overall Improvement Rating and on the Participant's Overall Self-Assessment Rating
Description: The proportion of participants rated as "improved" comprises those with complete remission, excellent, marked, or moderate improvement according to the Investigator's Overall Improvement Rating and those with excellent, good, or fair improvement the Participant's Overall Self-Assessment Rating. No improvement or deterioration (worsening of disease signs and symptoms compared to Baseline in the view of investigator/subject) comprise "not improved" status.
Time Frame: At Cycle 6 (Day 15±3 days of Treatment Cycle 6, 28 days per cycle)
Population: FAS (due to missing data number of participants differs from number at Baseline)
Measure: Number; unit: Percentage of participants
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Number analyzed (Participants) | 79 | 73
Percentage of participants
  Investigator | 93.7 | 78.1
  Participant | 94.9 | 84.9

ADVERSE EVENTS:
Arm/Group | EE20/Drospirenone (YAZ, BAY86-5300) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/86
Other Adverse Events (participants affected / at risk) | 34/87 | 19/86
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EE20/Drospirenone (YAZ, BAY86-5300) (N=87) | Placebo (N=86)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cervicitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Papilloma viral infection (Infections and infestations) | 0 | 1
Blood cholesterol increased (Investigations) | 3 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 0 | 1
White blood cells urine positive (Investigations) | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 2 | 2
Breast pain (Reproductive system and breast disorders) | 1 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 2
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0
Hypomenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 7 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 7 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less